CLINICAL TRIAL: NCT07218705
Title: A Prospective Study of Magnetocardiography for Disease Detection and Monitoring Treatment Outcomes in Amyloidosis
Brief Title: A Study Of MCG In Cardiac Amyloidosis
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mohamad Adnan Alkhouli, Principal Investigator, Mayo Clinic
Other Study IDs: 25-005053
Record Dates: First submitted 2025-10-16; First posted 2025-10-20 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Amyloidosis
MeSH Terms: conditions — Amyloidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with amyloidosis
  Interventions: Device: SandboxAQ CardiAQ Magnetocardiography

INTERVENTIONS:
Device: SandboxAQ CardiAQ Magnetocardiography — Magnetocardiography is a non-invasive, radiation-free imaging technique that detects the magnetic field generated by the electrical activity of the heart.

SUMMARY:
The primary objective of this observational study is to evaluate the utility of magnetocardiography (MCG) in diagnosing and monitoring disease progression in patients with amyloidosis, and to assess its effectiveness in comparison to other modalities, such as ECG.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥ 18 years on the date of consent
2. Ability for participant to comply with study requirements
3. Written informed consent

Exclusion Criteria

1. Pregnant or breastfeeding
2. Having an active atrial fibrillation episode as seen on most current 12-lead ECG
3. Active thoracic metal implants (including pacemaker, insertable cardiac monitor, or internal defibrillator).
4. External electrical pads or devices (e.g. Pacer pads, ECG electrodes, heart rate patch), that must remain on patient's chest during MCG scan
5. Inability to lie down in a supine/inclined position and stay still on the examination bed
6. Clinical conditions that in the opinion of the Investigator would compromise the safety of the patient or ability to complete the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study candidates may be identified and recruited in one of the following ways:
  * Amyloid Clinic (or other cardiology specialty clinics)
  * In-patient service at the study institution.
  * From the Principal Investigator or Co-Investigator clinical practices
  * Referral from other hospitals
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-12-03 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Receiver Operating Characteristic (ROC) curve | Baseline, 6 Months, 12 Months, 18 Months
  Receiver Operating Characteristic (ROC) curve is used to compare true positive rate vs false positive rate. This will be used to determine the sensitivity, specificity, and overall effectiveness of MCG.
Area Under the Curve (AUC) Magnetocardiography | Baseline, 6 Months, 12 Months, 18 Months
  Area Under the Curve (AUC) will be measured by mg*h/L.
Area Under the Curve (AUC) Electrocardiogram | Baseline, 6 Months, 12 Months, 18 Months
  Area Under the Curve (AUC) will be measured by mg*h/L.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad Alkhouli, M.D., M.B.A., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No